CLINICAL TRIAL: NCT05694520
Title: A Pragmatic Randomized Controlled Trial of Health Impact of Pistachios on Women
Brief Title: A Pragmatic Randomized Controlled Trial of Health Impact of Pistachios on Women With Gestational Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wei Chen, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDM trial
Record Dates: First submitted 2022-12-29; First posted 2023-01-23 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy

STUDY DESIGN:
Intervention Model Description: All subjects will be randomly assigned to intervention group (IG) or stand care control group (CG)), in an allocation ratio of (1:1) in blocks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stand care control group (CG) (No Intervention): According to the Chinese nutritional guidelines for GDM women, the energy intake of 1500-1800 kcal/d will be recommended for the included participants, who all have the pregestational BMI≥24 kg/m2. Standard care and a balanced diet will be recommended to the women in CG incorporating nuts intake of less than 2.5 oz per week.
- Intervention group (IG) (Experimental): The participants in the IG will be offered the otherwise same diet as their counterparts in the CG, except for the extra intake of pistachios of 1.5 oz thrice per week.
  Interventions: Other: pistachios consumption of 1.5 oz thrice per week

INTERVENTIONS:
Other: pistachios consumption of 1.5 oz thrice per week — According to the Chinese nutritional guidelines for GDM women, the energy intake of 1500-1800 kcal/d will be recommended for all the included participants with pregestational BMI≥24 kg/m2. Standard care and a balanced diet will be recommended to the women in CG incorporating the total nuts intake of less than 2.5 oz per week). While the women in the IG will be offered the otherwise same diet as their counterparts in the CG, except for the extra intake of pistachios of 1.5 oz thrice per week.
  Arms: Intervention group (IG)

SUMMARY:
Gestational diabetes mellitus (GDM) is the hyperglycemia with first onset or recognition during pregnancy, of which prevalence has been sharply increased worldwide in the past decades. Nuts offer numerous health benefits, mainly in relation to cardiovascular diseases as well as other chronic conditions. Pistachios have a balanced nutrition profile with lower fat [polyunsaturated fatty acids (PUFAs) and monounsaturated fatty acids (MUFAs)], higher protein, fiber (both soluble and insoluble), potassium, phytosterols, γ-tocopherol, vitamin K, xanthophyll carotenoids and rich antioxidant phytochemical constituents (stigmasterol, campesterol, resveratrol, catechins, lutein and zeaxanthin). Recent researches have found that nutritional intervention of the Mediterranean diet with an enhanced consumption of extra virgin olive oil and pistachios lowered incidence of GDM and other adverse outcomes (urinary tract infections, emergency C-sections, perineal trauma, large-for-gestational-age and small-for gestational age newborns) for pregnant women. Another clinical trial compared the acute metabolic effect of pistachios and isocaloric whole-wheat bread in women with GDM, finding significantly improved glucose and insulin responses, higher GLP-1 and lower gastric inhibitory polypeptide (GIP) levels in those consuming pistachios. However, more compelling evidences are still in need to throw light on the long-term effects of pistachio consumption on maternal and offspring's outcomes for GDM patients. Besides, effects of pistachios on the thorough metabolic profile of GDM patients also need to be elucidated.

This study aims to further demonstrate the long-term health effects of pistachio consumption on glycemic control, lipid profile, gut hormone responses, inflammatory condition and pregnancy outcomes for women with GDM.

The clinical study is a randomized, controlled, two-arm, parallel trial from the diagnosis of gestational diabetes to delivery consisting of six study visits including screening/consent. A total of 80 singleton pregnant women with confirmed diagnosis of GDM will be consecutively recruited, all with the pregestational body mass index (BMI) greater than 24 kg/m2. All subjects will be randomly assigned to intervention group (IG) or stand care control group (CG)), in an allocation ratio of (1:1) in blocks.

According to the Chinese nutritional guidelines for GDM women, the energy intake of 1500-1800 kcal/d will be recommended for the included women with pregestational BMI≥24 kg/m2. Standard care and a balanced diet will be recommended to the women in CG incorporating the total nuts intake of less than 2.5 oz per week). While the women in the IG will be offered the otherwise same diet as their counterparts in the CG, except for the extra intake of pistachios of 1.5 oz thrice per week. All participants will be followed up in 2 weeks initially and then once every 4-6 weeks until delivery or termination of pregnancy. The effect of different interventions on the glycemic profile (the continuous glucose monitoring (CGM) plus self-monitoring), lipid profile, gut hormone responses, inflammatory factors and metabolomics profiling (multi-omics data) will be monitored and compared. The pregnant outcome of the two groups will be also followed up and compared eventually.

With all data reviewed and analyzed, this study will add evidence to the long-term health effect of pistachios on GDM women.

ELIGIBILITY:
Inclusion Criteria:

* Chinese women at the age of 20-45 years, with Han ethnicity and singleton pregnancies
* Women who are at 20-30 weeks' singleton gestation and have the first onset of hyperglycemia which fulfills at least one of the following criteria: fasting glucose ≥5.1 mmol/L, 1 h glucose ≥10 mmol/L or 2 h glucose ≥8.5 mmol/L during the 2 h 75 g OGTT.
* Pregestational BMI greater than 24 kg/m2.
* Willing to comply with the research requirements

Exclusion Criteria:

* Gastrointestinal malabsorption and chronic diseases that alter nutrient metabolism
* Allergy or intolerance to pistachios
* Pre-existing diabetes, insulin resistance, impaired fasting glucose or impaired glucose tolerance
* Pregnancy with more than one fetus
* Current or planned corticosteroid therapy
* Current or planned beta adrenergic therapy
* Chronic medical conditions such as HIV/AIDS, kidney disease, or congenital heart disease
* Hematologic or autoimmune disease such as sickle cell disease, other hemoglobinopathies, lupus, or antiphospholipid syndrome

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-10 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-02-22 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Blood glucose response at 2 months | up to 2 months
  Change from baseline of the blood glucose response (time-in-range (TIR) on CGM, Hgb A1c, area under the curve of postprandial blood glucose (CGM)) after the nutritional management over 2 months
The incidences of adverse maternofetal outcomes | From date of intervention until the date of the delivery or termination of pregnancy, up to 4 months..
  The incidences of adverse maternofetal outcomes: emergency caesarean section (C-section), perineal trauma, pregnancy-induced hypertension and preeclampsia, prematurity, large-for-gestational age, and small-for-gestational age.

SECONDARY OUTCOMES:
Change from baseline the lipid profile at 2 months | up to 2 months
  Change from baseline of the lipid profile (TG, TC, HDL-C, LDL-C) after the nutritional management over 2 months
Change from baseline the inflammatory factors at 2 months | up to 2 months
  Change from baseline of the inflammatory factors (IL-6, hsCRP) after the nutritional management over 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China